CLINICAL TRIAL: NCT06073132
Title: An International, Multicenter, Randomized, Double-Blind, Parallel Group, Vehicle-Controlled, Phase 2/3 Study With Open-Label Extension Evaluating the Efficacy and Safety of Diacerein 1% Ointment for the Treatment of Generalized Epidermolysis Bullosa Simplex (EBS) [EBShield Study]
Brief Title: An International, Multicenter, Randomized, Double-Blind, Parallel Group, Vehicle-Controlled, Phase 2/3 Study With Open-Label Extension Evaluating the Efficacy and Safety of Diacerein 1% Ointment for the Treatment of Generalized Epidermolysis Bullosa Simplex (EBS)
Acronym: EBShield
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: TWi Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-203-EBS-007
Record Dates: First submitted 2023-09-12; First posted 2023-10-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Generalized Epidermolysis Bullosa Simplex
Keywords: Epidermolysis Bullosa Simplex; EBS
MeSH Terms: conditions — Epidermolysis Bullosa Simplex | interventions — diacerein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A AC-203 (Experimental): Double-blind, AC-203 Diacerein 1% ointment, QD
  Interventions: Drug: AC-203
- Part A Vehicle ointment (Placebo Comparator): Double-blind, Vehicle ointment, QD
  Interventions: Drug: Vehicle
- Part B AC-203 (Experimental): Open-label extension phase, AC-203 Diacerein 1% ointment, QD
  Interventions: Drug: AC-203

INTERVENTIONS:
Drug: AC-203 — The investigational product is formulated as 1% topical ointment
  Arms: Part A AC-203; Part B AC-203
Drug: Vehicle — Vehicle-only control study medication is the same formulation as investigational product without active ingredient
  Arms: Part A Vehicle ointment

SUMMARY:
The proposed Phase 2/3 trial with double-blind and open-label extension phases is an international, multicenter study designed to assess the efficacy and safety of diacerein 1% ointment in patients with generalized EBS.

DETAILED DESCRIPTION:
Epidermolysis bullosa simplex (EBS) is a genetic skin disorder characterized by skin fragility and recurrent blister formation, primarily caused by mutations in keratins 5 and 14. EBS has 3 common subtypes based on clinical severity and manifestations: localized EBS, intermediate EBS and severe EBS. Severe EBS and intermediate EBS collectively are also known as generalized EBS due to widespread blistering.

Disruption of the keratin 5/14 filament network in basal keratinocytes is a key factor in EBS pathogenesis, compromising skin integrity. The severity of EBS is linked to the extent of keratin mutations disrupting this network, particularly resulting in keratin aggregates in severe cases. Recent studies suggest that mutated keratin proteins can trigger inflammation, exacerbating EBS. Elevated proinflammatory cytokines, like IL-1β and IL-6, are observed in EBS patients, and IFN-γ may mediate inflammation, promoting keratin aggregations. As a result, targeting inflammation is considered a potential therapeutic approach in EBS.

AC-203 (diacerein 1% ointment) is a topical formulation of diacerein, well-known for its ability to inhibit IL-1β and other proinflammatory cytokines. Moreover, diacerein and its active metabolite, rhein, have demonstrated ability in reducing keratin aggregates in keratinocytes derived from severe EBS. Taken together, with its anti-inflammatory property and ability to diminish keratin aggregation, AC-203 shows promise in reducing the clinical severity of EBS.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 6 months old at Visit 2 (Day 1/Baseline A).
2. Patients has been clinically diagnosed with severe EBS or intermediate EBS, confirmed by documented genetic diagnosis to have autosomal dominant mutations in KRT5 or KRT14 gene.
3. Patient with ≥ 3% BSA of EBS lesions excluding palms and soles at Visit 2 (Day 1/Baseline A).
4. Patient's EBS lesions within the Treatment Area have an IGA score of ≥3 at Visit 2 (Day 1/Baseline A).
5. Patient/caregiver agrees to follow study medication application instructions.
6. Patient (and caregiver/legal guardian) agrees to report use of all prescription and over-the-counter medications, including topical therapies applied to the body, e.g., medical cleansers, bleach cleansers, bleach baths, topical antiseptics, topical disinfectants, etc. for the duration of the study.
7. Patient (and caregiver/legal guardian) is willing and able to comply with all study visits and all the protocol requirements, including completing questionnaires.
8. Patient (and caregiver/legal guardian) is able to provide written informed consent; assent based on age.
9. Female patient of childbearing potential must have a negative pregnancy test prior to randomization.
10. Female patient of childbearing potential is willing to practice highly effective contraception (i.e., pregnancy prevention method with a failure rate of < 1% per year) from Screening throughout the end of the study.

Exclusion Criteria:

1. Patient has a clinically significant skin disease other than EBS (e.g., psoriasis, atopic dermatitis, eczema, sun damage, etc.), or a vascular disorder associated with cutaneous erosions/ulcerations, that may confound assessments of efficacy or safety.
2. Patient has a clinically significant underlying medical condition, psychiatric condition (such as major depressive or psychotic disorder, severe intellectual disability, or alcohol or drug use disorder), or requires concomitant medication that based on the investigator's judgement may impair evaluation of the Treatment Area or exposes the patient to an unacceptable risk by study participation.
3. Patient has used any diacerein-containing product within 6 months prior to Visit 2 (Day 1/Baseline A).
4. Patient has had a cutaneous infection in the Treatment Area or use systemic antibiotics within 7 days prior to Visit 2 (Day 1/Baseline A).
5. Patient has uncontrolled diabetes mellitus (HbA1c ≥ 6.5%), hepatic enzyme abnormalities (alanine aminotransferase or aspartate aminotransferase >2.5 the upper limit of normal (ULN), or total bilirubin >2.0x ULN), or renal abnormalities (estimated glomerular filtration rate [eGFR]< 30 ml/min/1.73 m2) during the Screening period.
6. Patient has a current malignancy, or a history of treatment for a malignancy within 5 years (with the exception of treated non-melanoma cutaneous malignancy e.g., surgically resected with clear margins) prior to Visit 2 (Day 1/Baseline A).
7. Patient is treated with protocol-excluded topical therapies other than steroids within 2 weeks prior to Visit 2 (Day 1/Baseline A) that might influence the assessment of the Treatment Area throughout the study period.
8. Patient has been treated with topical steroids on the EBS lesions within 2 weeks or systemic steroids within 4 weeks. prior to Visit 2 (Day 1/Baseline A). (Note: inhaled and ophthalmic products containing steroids are allowed.)
9. Patient has been treated with: (a) an approved biologic anti-inflammatory therapy (such as monoclonal antibodies that target to modulate the immune responses) and (b) other immunosuppressive/immunomodulatory therapies or chemotherapy within 8 weeks prior to Visit 2 (Day 1/Baseline A).
10. Patient has been treated with any investigational drug or device within 30 days or 5 half-lives, whichever is longer, prior to Visit 2 (Day 1/Baseline A).
11. Patient has a history of allergy or hypersensitivity to any component of study medications, including diacerein or rhein.
12. Patient is pregnant or breastfeeding/lactating.
13. Patient has a planned or anticipated major surgical procedure or other activity that would interfere with their ability to comply with protocol requirements.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving treatment success on the IGA of the Treatment Area, in which treatment success is defined as a score of 0 or 1 with at least a 2-point reduction | from Baseline A (Visit 2/Day 1) to Week 8 (Visit 5/EOT)
  The static IGA is the investigator's visual clinical assessment of the average overall intensity of lesions in the designated Treatment Area at a particular time point. EBS-IGA is a 5-point scale is a 5-point scale (clear=0; almost clear=1; mild=2; moderate=3; severe=4)

SECONDARY OUTCOMES:
Change in % BSA of EBS lesions in the Treatment Area | from Baseline A (Visit 2/Day 1) to Week 8 (Visit 5/EOT)
  The Body Surface Area (BSA) of the Assessment Area will be collected for all lesions included within the Treatment Area using the palmar method
Change in pain intensity score | Baseline A (Visit 2/Day 1) to Week 8 (Visit 5/EOT)
  Wong-Baker FACES® Pain Rating Scale will be used for patients 3 years and older.
Change in pruritus intensity score | from Baseline A (Visit 2/Day 1) to Week 8 (Visit 5/EOT)
  ItchyQuant will be used for patients aged 6 years and older, including adult patients
Change in EBDASI score (skin activity) | from Baseline A (Visit 2/Day 1) to Week 8 (Visit 5/EOT).
  The EBDASI is a valid and reliable EB-specific outcome measurement tool to assess the overall extent of disease activity and damage in patients with various subtypes of EB, including EBS. Section I (skin), the severity of disease, including erosion/blisters/crusting etc., will be measured at 12 different skin sites.
Change in the QOLEB score | from Baseline A (Visit 2/Day 1) to Week 8 (Visit 5/EOT)
  The Life Epidermolysis Bullosa (QOLEB) questionnaire is a valid and reliable, EB-specific QOL measurement tool, for the quantification of QOL in patients with various subtypes of EB, including EBS. It consists of 17 questions with four response choices from "not at all" to "constant"

CONTACTS AND LOCATIONS:
Locations (36):
- United States (9):
  - Mission dermatology Center, Rancho Santa Margarita, California
  - Stanford University, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Pediatric Skin Research, LLC, Miami, Florida
  - Northwestern University - Lurie Childrens's Hospital, Chicago, Illinois
  - Stony Brook Dermatology, Stony Brook, New York
  - Cincinnati Childrens Hospital, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
- Australia (3):
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Premier Specialists, Kogarah
  - Sydney Children's Hospital, Randwick
- Universitaetsklinik fuer Dermatologie und Allergologie, Salzburg, Austria
- UZ Leuven, Leuven, Belgium
- Hopital Necker-Enfants Malades, Paris, France
- Greece (2):
  - Andreas Syggros Hospital 1st University Clinic of Skin and Venereal Diseases of Athens, Athens
  - Hospital of Skin and Venereal Diseases of Thessaloniki, Thessaloniki
- Postgraduate Institute of Medical Education and Research (PGIMER), Chandigarh, India
- Children's Health Ireland, Dublin, Ireland
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Italy (5):
  - IRCCS, AOUBO, Policlinico Sant'Orsola, Bologna
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico Milano, Milan
  - Università degli Studi di Modena e Reggio Emilia (UNIMORE), Modena
  - Istituto Dermopatico dell'Immacolata (IDI) - Istituto di, Rome
  - UOS "Centro delle Dermatosi Croniche Complesse e Genodermatosi" UOC Dermatologia, Rome
- Hospital Tunku Azizah (Hospital Wanita Dan Kanak-kanak Kuala Lumpur), Kuala Lumpur, Malaysia
- Philippines (3):
  - Asian Hospital, City of Muntinlupa
  - Iloilo Doctors Hospital, Iloilo City
  - Health Cube Medical Clinics, Mandaluyong
- OT.CO Clinic Osipowicz & Turkowski, Warsaw, Poland
- Gangnam Severane Hospital, Seoul, South Korea
- Hospital Universitario La Paz, Madrid, Spain
- National Cheng Kung University Hospital, Tainan, Taiwan
- Sheikh Khalifa Medical City (SKMC), Abu Dhabi, United Arab Emirates
- United Kingdom (2):
  - Great Ormond Street Hospital (GOSH) for Children NHS Foundation Trust - Somers Clinical Research Facility (CRF), London
  - University Hospitals Birmingham NHS Foundation Trust (UHB), Solihull

IPD SHARING:
Plan to Share IPD: No